CLINICAL TRIAL: NCT03363932
Title: French Observatory of Congenital Ventricular Septal Defect With Pulmonary Overload
Acronym: FRANCISCO
Status: Active, not recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 17.10.55
Record Dates: First submitted 2017-11-21; First posted 2017-12-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease
Keywords: Ventricular septal defect; Congenital heart disease; Outcome
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perimembranous VSD with high pulmonary flow rate: It is an observational study, no intervention or examination will be realized for the sole purpose of the study. Patient management will be at the discretion of referral cardiologists according to the practices of the centers.
  As part of the usual follow-up of these patients, the participating centers collect the clinical and echocardiography data from inclusion and the following year, as well as data from a functional assessment at baseline and at one year. and the collection of cardiovascular events at 5 years and 10 years of follow-up.
  Data from a possible percutaneous or surgical closure procedure will be collected. The indication of VSD closure will be left to the discretion of participating centers. There will be no recommendation for percutaneous or surgical closure of VSD for the sole purpose of this observatory.

SUMMARY:
Ventricular septal defects (VSD) are the most common cardiac congenital heart defect (about 1/3 of patients with congenital heart disease). VSD management is related to hemodynamics and anatomical localization and the occurrence of complications. Small perimembranous VSD without pulmonary hypertension and without significant left to right shunting are tolerated, whereas large VSD with pulmonary hypertension require early surgical management in the first months of life. The management uncertainties concern the medium-sized perimembranous VSD causing a significant left-right shunt but without pulmonary hypertension, which are of variable treatment (surgical correction, percutaneous treatment, medical or abstention). There are no recommendations or consensus on the preferred indication of a therapeutic attitude.

The Pediatric and Congenital Cardiology Subsidiary, within the French Society of Cardiology, set up an observatory of perimembranous VSD with significant shunting, without pulmonary hypertension the objectives of this study are:

* To study the incidence of cardiovascular events in perimembranous VSD and search for predictive anatomical markers of events.
* To study the evolution of echocardiographic and functional data of patients having percutaneous or surgical closure compared to patient managed medically.

This observatory will provide a better understanding of the therapeutic algorithm in the management of VSD with pulmonary overload without pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 1 year old
* Having a perimembranous VSD with pulmonary overload defined by "a left-right shunt and a z-score of the left ventricular end-diastolic diameter> = 2".
* Consent for inclusion in the study was signed by the parents or legal guardian for minors, by the patient for the adults.

Exclusion Criteria:

* Congenital heart disease associated with membranous VSD
* Stenosis of the left ventricular outflow tract (average gradient ≥20 mmHg)
* Aortic insufficiency
* sub-pulmonary stenosis (mean gradient ≥20 mmHg)
* Tricuspid insufficiency ≥ 2/4
* History of cardiac surgery or cardiac interventional catheterization
* Shunt right-left through the VSD
* Pulmonary Arterial Hypertension defined on the data of a catheterization by PAPM> = 25 mmHg and pulmonary vascular resistance> = 3 UW.m²
* Active infectious endocarditis
* Cardiac insufficiency according to the "ESC 2016" criteria, other than a symptomatology of pulmonary hyper flow during the first year of life. Heart failure is defined by the presence of clinical signs of heart failure associated with a structural or cardiac functional abnormality resulting in a decrease in cardiac output and / or an increase in filling pressures.
* History of persistent or chronic atrial arrhythmia (atrial flutter, atrial tachycardia or chronic atrial fibrillation or requiring electrical cardioversion, drug therapy or endocavitary ablation)
* History of sustained ventricular arrhythmia (duration> = 30 seconds)
* Complete BAV
* Refusal of the patient or guardian to participate in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who agreed to participate in the study, met the inclusion criteria, and treated in a French medical and surgical center with pediatric and congenital cardiology activity
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Cardiovascular Events at 5 Years of Perimembranous VSD with pulmonary overload | 5 years of follow-up
  The main criterion "cardiovascular event" is a composite criterion. At least 1 of the following criteria is required for the primary criterion to be met:
  * endocarditis,
  * aortic stenosis (mean gradient> 20 mmHg)
  * aortic insufficiency
  * left ventricular outflow tract stenosis (mean gradient> 20 mmHg)
  * tricuspid insufficiency ≥2
  * surgery or cardiac interventional catheterization for an abnormality in relation to the VSD (other than simple closing)
  * persistent supraventricular arrhythmias, sustained ventricular arrhythmia,
  * stroke
  * Complete atrioventricular block (AVB)
  * Pulmonary Arterial Hypertension (PAH)
  * heart failure
  * cardiovascular deaths,
  * severe haemolysis (= requiring transfusion or interventional catheterization or surgical).

SECONDARY OUTCOMES:
Anatomical predictive elements of events at 5 years of follow-up. | 5 years of follow-up
  The event criterion meets the same definition as the primary judgment criterion. The association between anatomical elements (size of the VSD, presence of aneurysm, diameter and depth of the aneurysm, septo-aortic angulation) and cardiovascular events will be studied.
Evolution of the left ventricular end diastolic diameter z-score one year after VSD closure | 1 year of follow-up
  Evolution of the left ventricular end diastolic diameter z-score one year after VSD closure
Incidence of cardiovascular events of "high-flow" VSDs according to the different therapeutic options at 5 years of follow-up | 5 years of follow-up
  Incidence of cardiovascular events of "high-flow" VSDs according to the different therapeutic options (medical - percutaneous closure - surgical closure) at 5 years of follow-up. The event criterion meets the same definition as the primary judgment criterion.
Incidence of cardiovascular events of "high-flow" VSDs according to the different therapeutic options at 10 years of follow-up. | 10 years of follow-up
  Incidence of cardiovascular events of "high-flow" VSDs according to the different therapeutic options (medical - percutaneous closure - surgical closure) at 10 years of follow-up. The event criterion meets the same definition as the primary judgment criterion.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Hopital Europeen Georges Pompidou, Paris
  - Gh Sud Hopital Haut Leveque, Pessac
  - Chu Toulouse - Hopital Des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penny DJ, Vick GW 3rd. Ventricular septal defect. Lancet. 2011 Mar 26;377(9771):1103-12. doi: 10.1016/S0140-6736(10)61339-6. Epub 2011 Feb 23. PMID 21349577
- [Background] Karonis T, Scognamiglio G, Babu-Narayan SV, Montanaro C, Uebing A, Diller GP, Alonso-Gonzalez R, Swan L, Dimopoulos K, Gatzoulis MA, Li W. Clinical course and potential complications of small ventricular septal defects in adulthood: Late development of left ventricular dysfunction justifies lifelong care. Int J Cardiol. 2016 Apr 1;208:102-6. doi: 10.1016/j.ijcard.2016.01.208. Epub 2016 Jan 23. PMID 26844920
- [Background] Videbaek J, Laursen HB, Olsen M, Hofsten DE, Johnsen SP. Long-Term Nationwide Follow-Up Study of Simple Congenital Heart Disease Diagnosed in Otherwise Healthy Children. Circulation. 2016 Feb 2;133(5):474-83. doi: 10.1161/CIRCULATIONAHA.115.017226. Epub 2015 Dec 18. PMID 26683488
- [Background] Odemis E, Saygi M, Guzeltas A, Tanidir IC, Ergul Y, Ozyilmaz I, Bakir I. Transcatheter closure of perimembranous ventricular septal defects using Nit-Occlud((R)) Le VSD coil: early and mid-term results. Pediatr Cardiol. 2014 Jun;35(5):817-23. doi: 10.1007/s00246-013-0860-8. Epub 2014 Jan 12. PMID 24413836
- [Background] Chungsomprasong P, Durongpisitkul K, Vijarnsorn C, Soongswang J, Le TP. The results of transcatheter closure of VSD using Amplatzer(R) device and Nit Occlud(R) Le coil. Catheter Cardiovasc Interv. 2011 Dec 1;78(7):1032-40. doi: 10.1002/ccd.23084. Epub 2011 Jun 6. PMID 21648053
- [Result] Guirgis L, Valdeolmillos E, Vaksmann G, Karsenty C, Houeijeh A, Hery E, Amedro P, Pangaud N, Benbrik N, Vastel C, Legendre A, Jalal Z, Hadeed K, Ladouceur M, Iserin L, Laux D, Iriart X, Warin Fresse K, Leobon B, Harchaoui S, Lambert V, Bonefoy R, Basquin A, Chalard A, Douchin S, Bouzguenda I, Denis C, Lucron H, Bosser G, Barre E, Urbina-Hiel B, Helms P, Ansquer H, Hauet Q, Leborgne AS, Cohen L, Lupoglazoff JM, Guirgis M, Gronier C, Maragnes P, Moceri P, Mauran P, Bertail C, Lefort B, Godart F, Baruteau AE, Ovaert C, Bonnet D, Combes N, Khraiche D, Houyel L, Thambo JB, Mostefa-Kara M, Hascoet S; FRANCISCO investigators. Cardiovascular events in perimembranous ventricular septal defect with left ventricular volume overload: a French prospective cohort study (FRANCISCO). Cardiol Young. 2021 Oct;31(10):1557-1562. doi: 10.1017/S1047951121002717. Epub 2021 Sep 23. PMID 34551835